CLINICAL TRIAL: NCT03813745
Title: Timing of COC Denudation and Embryo Quality: A Prospective Randomised Sibling-Oocyte Study
Brief Title: Timing of COC Denudation and Embryo Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Elif Esra Uyar, Medical Doctor, Acıbadem Atunizade Hospital
Other Study IDs: COCdenudation
Record Dates: First submitted 2019-01-10; First posted 2019-01-23 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-01

CONDITIONS: Infertility, Female
Keywords: embryo quality; denudation; IVF; ICSI
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early denudation: Cumulus-oocyte complexes will be denudated in 30 min after oocyte retrieval
  Interventions: Other: early denudation
- late denudation: Denudation will be done 2 hr after oocyte retrieval
  Interventions: Other: late denudation

INTERVENTIONS:
Other: early denudation — COCs will be denudated in 30 min after oocyte retrieval
  Groups: early denudation
Other: late denudation — COCs will be denudated 2 hr after oocyte retrieval
  Groups: late denudation

SUMMARY:
The relation between the timing of COC denudation and oocyte /embryo quality is controversial. The aim of this study is to examine whether timing of denudation of sibling oocytes has any effect on embryo quality.

DETAILED DESCRIPTION:
Retrieved sibling cumulus-oocyte complexes (COCs) will be randomly divided into two groups, in the first group denudation will be in 30 minutes after oocyte retrieval, in second group denudation will take place after 2 hours of incubation.

ELIGIBILITY:
Inclusion Criteria:

* COH with GnRH antagonist cycle
* 5 or more oocytes collected

Exclusion Criteria:

* Fewer than 4 oocytes after retrieval
* Previous history of total fertilization failure or oocyte maturation arrest
* Male partner requiring surgical sperm retrieval (MESA or TESA).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Those infertile patients eligible for the study design who are planned to be treated with microinjection and has given written informed consent
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-25 (Estimated)

PRIMARY OUTCOMES:
Number of good quality cleavage embryos | 3 days after microinjection
  Quality of embryos will be assessed morphologically on day 3
Embryo utilization rate | 1 week after microinjection
  Embryo utilization rate is defined as the number of embryos utilized (transferred or cryopreserved) per number of 2PN zygotes.

SECONDARY OUTCOMES:
Fertilization rate | 16-18 hour after microinjection
  Proportion of injected oocytes with 2PN the day after injection
Cleavage rate | 2 days after microinjection
  Proportion of cleaved zygotes on day 2
Blastulation rate | 1 week after microinjection
  Blastocyst rate per oocyte

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Altunizade Hospitai, Istanbul, Turkey (Türkiye)